CLINICAL TRIAL: NCT01304199
Title: Cancer Survivorship Issues: A Survey of Patients in India.AIIMS Study (CANSURVIVE)
Acronym: CANSURVIVE
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: All India Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Bidhu Kalyan Mohanti, Professor Department of Radiation Oncology, All India Institute of Medical Sciences
Other Study IDs: IEC/NP-252/2010
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-07

CONDITIONS: Cancer
Keywords: Cancer survivor; Neoplasms; Treatments; Physical status; Psychosocial status; Survivorship survey; Survivorship care; Research; Cancer patient
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adult Cancer Survivors: Intervention:
  Behavioural:
  Questionnaires for patient/family caregiver interview

SUMMARY:
The purpose of this study is to assess the various aspects of life in the cancer survivors in India. Cancer survivor is defined as "an individual diagnosed with cancer and who has survived the disease and treatment, and for the rest of his/her life".

Cancer survivors are at increased risk of developing various physical and psychosocial conditions, which require to be identified and attended within the cancer care system.

Survivorship research is seen as addressing the medical, functional, and health related issues of individuals diagnosed with cancer, as well as that of their families.

DETAILED DESCRIPTION:
It is estimated that approximately 25 million people are living as cancer survivors worldwide. The cancer survivors are those individuals who live beyond a cancer diagnosis and its therapy. Within the existing health care system, the cancer care models are largely focused on diagnostic methods, treatment aspects, cure, and disease failure and survival rates. There is very little research and intervention approaches for the after-effects of cancer diagnosis and treatments for an individual cancer patient. Cancer survivors are at increased risk of developing various physical and psychosocial conditions, which require to be identified and attended within the cancer care system. In the developing countries like India, the cancer cure rates are improving due to improvements in comprehensive diagnostic and treatment strategies. Cancer survivorship research will be valuable to enhance our understanding and care approaches to these vulnerable individuals in our society. There is lack of evaluation tools which can completely fit to assess all issues such as physical, social, financial, mental aspects of a cancer survivor.

Hence the investigators of this observational study have prepared an empirical cancer survivorship questionnaire (CSQ) which will document the patient's disease and treatment details and obtain subjective responses from the patient(and/or family care giver) related to the physical, functional, social, economic and mental aspects of daily living of a cancer survivor. In order to assess the mental status of the survivors, the investigators have also included the widely used and internationally accepted MINI (Mini-international neuropsychiatry interview) version along with the CSQ in this survey. Researchers and clinicians working in non-profit and academic setting such as this institution are allowed to make copies of this MINI questionnaire for the purpose of clinical and research use. For the present study, MINI version is suitably modified to exclude the items which are already in the CSQ, and certain items are reframed for the socio-cultural requirement. Both the CSQ (45 items) and MINI-modified (13 items) will be applied simultaneously in this survey as a direct face to face response documentation from the patient (cancer survivor), along with his/her family member. Patients will be chosen for this cross-sectional survey during the follow-up visit to a cancer clinic of this hospital, at least 3 months after the completion of cancer diagnosis and therapy. Each participant is expected to complete the survey at the first encounter, however, a provision is made to report any missing information at later visit.

An interim analysis will be carried out after the survey of first 50 patients to observe the trends in the findings. However, this will not impact the further accrual, except for making some changes in the survey parameters if at all needed.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were treated with curative intent and are on hospital follow up visit.
* Patients aged above 18 years and of both sexes.
* Patients who have no evidence of disease at the time of collecting information.
* Patients or family carers who are able to comprehend and communicate.
* Cancer diagnosed and treated at AIIMS, at least 3 months before entry into the study.

Exclusion Criteria:

* Patients who refuse to provide informed consent for this study.
* Patients treated for cancer outside AIIMS.
* Patients who have recurrence or disease failure for which they are or are not receiving salvage therapy.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study will evaluate the cancer patients visiting Dr BRAIRCH,AIIMS,New Delhi,India after a cancer diagnosis and the cancer treatments have been completed.
  The patients will be entered into this study(survey) during the follow up visits to the clinic.
  Patients will be evaluated and assessed for their cancer survivorship issues on the basis of a questionnaire (CSQ) developed by the investigators after the literature review. The mental status of the survivors is assessed by a MINI- international neuro-psychiatric interview, suitably modified to incorporate the CSQ in this survey.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2013-07 (Estimated); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
To study the cancer survivorship experience(as binary responses) | 1 year
  Behavioral: Questionnaires and medical records. The cancer survivors' physical, social, economic and psychological issues will be assessed as verbal response.The survey questionnaires will document the sequelae of cancer and its treatment during the face to face interview and by collecting information from the individual cancer survivor's medical records
To assess the mental status of cancer survivors | 1 year
  Behavioral:MINI-international neuro-psychiatric questionnaire(modified for local use)

SECONDARY OUTCOMES:
To identify the differences if any, in the cancer survivorship issues by age(Less than 50 or greater than 50 years) | up to 6 months after patient accrual
  This cancer survivorship survey will include adult cancer survivors post-therapy. Survivors of various neoplasms will be accrued for this survey.
To define follow up care for cancer survivors in India. | up to 6 months after patient accrual
  This survey of 200 adult cancer survivors will analyse various issues-physical, social, psychological and economic which adversely impact the life of cancer survivors in India.
  This analysis will help in evolving a feasible approach towards implementation of follow up care practice for cancer survivors.

CONTACTS AND LOCATIONS:
Overall Officials: BIDHU K MOHANTI, MD, Study Chair — All India Institute of Medical Sciences; Jaspreet Kaur, MD, Study Director — All India Institute of Medical Sciences; Sudhir K Khandelwal, MD, Study Director — All India Institute of Medical Sciences; Ravindra M Pandey, PhD, Study Director — All India Institute of Medical Sciences
Locations (1):
- All India Institute of Medical Sciences Dr.B.R.A.Institute Rotary Cancer Hospital, New Delhi, National Capital Territory of Delhi, India

REFERENCES:
- [Derived] Mohanti BK, Kaur J. Living experiences of Indian adult cancer survivors--a brief report. Asian Pac J Cancer Prev. 2015;16(2):507-12. doi: 10.7314/apjcp.2015.16.2.507. PMID 25684479
- See also: Office of Cancer Survivorship CCPS, Cancer Control & Population Sciences.National Cancer Institute 6130 Executive Boulevard Room 6134 Executive Plaza North Rockville, Maryland 20852 Phone: 301-594-6776 Fax: 301-594-6787 — http://cancercontrol.cancer.gov/ocs/